CLINICAL TRIAL: NCT02118298
Title: Allocentric Memory as a Novel Measure of Cognitive Inefficiency: Sensitivity in Multiple Sclerosis (MS) Subjects and Relationship With Resting State Functional MRI
Brief Title: Allocentric Memory in MS and Resting State Functional MRI
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1401013272
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: Ages 18 - 66, 10 years or less of MS,
- Demographically matched controls: Ages 18 - 66, No known neurological disorder, no learning disorder, and no psychiatric disturbance that is actually interfering with life.

SUMMARY:
The goals of this study are to 1. Investigate the sensitivity of allocentric visual memory when compared to more established measures of cognition in identifying cognitive difficulties among MS subjects when compared to controls. 2. Determine which cognitive test variable will be most strongly associated with self and informant reports of cognition. 3. Determine which MRI metric will be most strongly related to neuropsychological test performance 4. Determine the degree to which allocentric visual memory is related to functional connectivity on fMRI.

DETAILED DESCRIPTION:
This is a cross-sectional, case-control, observational experimental design. The study will enroll subjects with multiple sclerosis (MS) and age/gender matched on a battery of neuropsychological cognitive tests and self-report measures of cognition.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Right handed
* Capacity to provide informed consent and sign consent
* Diagnosis of Relapsing Remitting MS that meets the revised McDonald Criteria (2010) within the last 10 years
* EDSS 0- 5.5

Exclusion Criteria:

* Diagnosis of primary progressive MS
* Contraindications for MRI
* Subjects required to take medications known to either benefit or adversely affect cognition at the time of testing and impact neuroimaging
* Non-MS neurological disorders
* Other medical or psychiatric disorders likely to affect cognitive performance
* Active immunodeficiency, chronic infections, or history or progressive multifocal leukoencephalopathy
* Individuals with severe level of depression on the BDI-II or severe anxiety on the BAI
* MS subjects who are actively experiencing acute exacerbation in symptoms and they must be at least 4 weeks free of steroid medication, are currently taking a chemotherapy agent, or have changed medication in the last two months
* Subjects who fail symptom validity measures during neuropsychological testing will be excluded

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with relapsing remitting Multiple Sclerosis and demographically matched controls will be recruited for this study. The MS subjects will consist of patients who were referred for a neuropsychological evaluation and neuroimaging as part of standard practice of care to evaluate for cognitive difficulties and/or track disease progression.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Minimal Assessment of Cognitive Function in MS (MACFIMS) | Baseline
  The MACFIMS is composed of seven neuropsychological tests, covering five cognitive domains commonly impaired in MS (processing speed/working memory, learning and memory, executive function, visual-spatial processing and word retrieval)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin C Brown, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided